CLINICAL TRIAL: NCT03717103
Title: A Phase 1 Study Evaluating the Safety, Tolerability, and Initial Efficacy of Recombinant Human Anti-cluster Differentiation Antigen 47 (CD47) Monoclonal Antibody Injection (IBI188) in Patients With Advanced Malignancies
Brief Title: A Phase 1 Study Evaluating the Safety, Tolerability, and Initial Efficacy of IBI188 in Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI188A101
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Advanced Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI188 (Experimental): Part A : Initial dose escalation, Part B : Maintenance dose escalation
  Interventions: Drug: IBI188

INTERVENTIONS:
Drug: IBI188 — Part A: 0.1 mg/kg IV QW, 0.3 mg/kg IV QW, 1 mg/kg IV QW. Part B: 1mg/kg IV D1+3, 10, 20, 30 mg/kg IV D8 QW or 45mg/kg D8 IV Q3W.
  Other Names: Letaplimab

SUMMARY:
This is an open-label, dose escalation, Phase I study to evaluate the safety, tolerability, pharmacokinetics and efficacy in patients with advanced malignancies.

DETAILED DESCRIPTION:
Phase Ia study is composed of two stages: Phase Ia Part A initial dose escalation and Phase Ia Part B maintenance dose escalation. Both parts will adopt the classical 3+3 dose escalation design. The starting dose for phase Ia part A is 0.1 mg/kg QW, followed by 2 dose cohorts (0.3 mg/kg QW and 1 mg/kg QW). Duration of dose limiting toxicity (DLT) observation is 14 days.

Phase Ia Part B will have 4 dose cohorts(3mg/kg QW#10mg/kg QW#20mg/kg QW #30mg/kg QW and 45mg/kg Q3W). DLT observation period is 28 days. The subject number for each cohort in Phase Ia Part B will be increased to 6 if the subject number enrolled in each cohort is less than 6

ELIGIBILITY:
Inclusion Criteria:

1. Advanced solid tumors and lymphomas defined by:

   * Histologically/cytologically confirmed solid tumors and lymphomas
   * Solid Tumors failed from standard therapy
   * Lymphoma patients who have had at least two standard treatment failures
2. Subject has at least 1 measurable disease per RECIST v1.1. Lymphomas have at least one measurable lesion and 18FDG-avid lesion according to the Lugano 2014 criteria.
3. Male or female subject above 18 years
4. ECOG Performance Status 0 to 1
5. Must have adequate organ and bone marrow function, including the following:

   * Blood routine: absolute neutrophil count (ANC) ≥ 1.5 x10^9/L; platelet count ≥ 75 x 10^9/L; hemoglobin ≥ 10 g/dL. (For subjects with AML, WBC < 25×10^9/L was required , and there is no restriction for the rest in blood routine test ).
   * Hepatic: total bilirubin ≤ 1.5 times of the upper limit of normal (ULN), aspartate transaminase (AST) and/or alanine aminotransferase (ALT) ≤ 2.5 X ULN (≤5 X ULN if with liver involvement). total bilirubin ≤ 3×ULN if subjects were diagnosed with Gilbert syndrome.
   * Renal: serum creatinine ≤ 1.5 X ULN or estimated creatinine clearance ≥50mL/min. Urinary protein < 2+. For subjects with urinary protein ≥2+ at baseline, a 24h urine collection should be performed with urine protein < 1g.
   * Coagulation tests INR < 1.5, partial prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN
6. Subjects with life expectancy of ≥ 12 weeks
7. Female subjects of child-bearing potential or male subjects with female partners of child-bearing potential must be willing to use viable contraception method that is deemed effective by the investigator throughout the treatment period and for at least 6 months following the last dose of study drug.
8. Be willing to sign the Informed Consent Form (ICF), and can follow the visit schedule and procedures defined in the protocol.

Exclusion Criteria:

1. Previous exposure to any anti-CD47 monoclonal antibody or SIRPα antibody.
2. Subjects participating in any other interventional clinical study
3. Received blood transfusion, biologic G-CSF, GM-CSF, erythropoietin, thrombopoietin (TPO) or IL-11within 3 weeks prior to the first dose of study drug
4. Receive the last dose of anti-tumor therapy (chemotherapy, endocrine therapy, targeted therapy, immunotherapy or tumor embolization, etc.) within 3 weeks before the first dose of the study.
5. Immunosuppressive drugs were used within 7 days before the first dose of the study
6. Plan to receive live attenuated vaccines within 4 weeks before the first dose treatment or during the study period.
7. Has undergone major surgery (craniotomy, thoracotomy or laparotomy) or is expected to require major surgery during the first dose of the study.
8. Any remaining AEs > grade 1 from prior anti-tumor treatment as per CTCAE v5.0, with exception of the residual hair loss nor fatigue
9. Had received total pelvic radiotherapy before.
10. Central nervous system metastases:
11. Subjects with active or suspected autoimmune disease or a history of the disease in the past two years
12. known history of primary immunodeficiency.
13. known history of active pulmonary tuberculosis.
14. known history of allograft transplantation and history of allogeneic hematopoietic stem cell transplantation.
15. known to be allergic to any IBI188 preparations.
16. Ascites of clinical significance, including any ascites that may be detected by physical examination, previously treated or still in need of treatment, may be enrolled if only a small amount of ascites is shown on imaging but asymptomatic.

18. Subjects with moderate bilateral pleural effusion, or massive pleural effusion on one side, or respiratory dysfunction requiring drainage.

19. Pregnant or nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs), Serious Adverse Events (SAE)Number of patients with AEs and SAEs | 24 months
  Incidence, correlation with the study drug and severity of all adverse events (AEs), treatment-emergent adverse events (TEAEs), adverse events of special interest (AESIs) and serious adverse events (SAEs).

SECONDARY OUTCOMES:
Preliminary anti-tumor activity of IBI188 (Objective Response Rate) | 24 months
  Objective Response Rate (ORR) is the percentage of Complete Response (CR) plus partial response (PR) assessed by RECIST v1.1 criteria for solid tumors and Lugano2014 criteria for lymphoma.
Pharmacokinetics: Cmax | 24 months
  Maximum concentration(Cmax) of the drug after administration
Pharmacokinetics: AUC | 24 months
  The area under the curve (AUC) of serum concentration of the drug after the administration.
Immunogenicity | 24 months
  Anti-Drug Antibodies (ADA) will be tested and percentage of ADA positive patients will be calculated to evaluate immunogenicity of IBI188.

CONTACTS AND LOCATIONS:
Overall Officials: Song Yuqin, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China